CLINICAL TRIAL: NCT06970496
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability and Preliminary Efficacy of B019 Injection in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma.
Brief Title: A Clinical Trial of B019 Injection in Patients With Relapsed or Refractory B-cell Non-Hodgkin's Lymphoma.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceutical Group Biological Therapy Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B019-102
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-05

CONDITIONS: Relapsed or Refractory B Cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B019 (Experimental)
  Interventions: Drug: B019

INTERVENTIONS:
Drug: B019 — B019： Intravenous infusion, 2.0×10^6 cell/kg-8.0×10^6 cell/kg

SUMMARY:
The purpose of the study is to evaluate the safety、tolerability and preliminary efficacy of B019 in subjects with relapsed or refractory B-cell non-Hodgkin's lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who can fully understand this trial and voluntarily sign the informed consent form (ICF) before any research-related procedures;
2. Histologically confirmed B-cell non-Hodgkin's lymphoma (B-NHL) with specified pathological subtypes;
3. Histologically confirmed CD19 and/or CD22 positivity;
4. Expected survival time exceeding 12 weeks;
5. ECOG performance status 0-1 (Ia) or 0-2 (Ib);
6. At least one measurable lesion in two dimensions according to the Lugano 2014 criteria;
7. Bone marrow, liver, kidney, and cardiac-pulmonary functions meeting the specified requirements; 8 Subjects who were evaluated by the researchers as tolerant to the collection of peripheral blood mononuclear cells (PBMC); 9 Subjects who were evaluated by the researchers as having no contraindications for lymphodepleting chemotherapy.

Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma; However, secondary CNS lymphoma without clinical symptoms can be enrolled after being determined by the researchers；
2. Use of the prescribed drugs or treatments within the specified time before the collection of PBMC;
3. Prior allogeneic hematopoietic stem cell transplantation;
4. Systemic intravenous infusion treatment or uncontrollable bacterial, fungal or viral infection within 2 weeks before signing the ICF;
5. A history of deep vein thrombosis or pulmonary embolism or anticoagulant therapy within 6 months before signing the ICF;
6. A clinically significant history of severe heart disease within 6 months before signing the ICF;
7. Terminal organ damage or autoimmune diseases requiring systemic immunosuppressive/systemic treatments within 2 years before signing the ICF; Or have graft-versus-host disease;
8. Prescribed malignant tumors within 5 years before signing the ICF;
9. Intestinal obstruction caused by tumor compression or vascular compression requiring emergency treatment; gastrointestinal involvement with a risk of bleeding assessed by the researchers;
10. Clinically significant CNS diseases in the past or at the time of screening;
11. A history of severe allergic reactions to the drugs or excipients that were definitely needed in this study. Or have a history of allergic reactions to tocilizumab;
12. Any indwelling tubes or drainage tubes in the bodies, the use of dedicated central venous access catheters is permitted;
13. Pregnant or breastfeeding women; or male or female subjects who are unwilling to use contraception from the time of signing the ICF until 1 year after receiving B019 injection cell infusion or until CAR is detectable in peripheral blood.;
14. The subjects who have participated in other clinical studies within the past 1 month, or whose last medication use for the last clinical study is still within the 5 half-life periods of the current drug at the time of screening;
15. Other circumstances that the researchers consider unsuitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Approximately 2 years
  Measurement of DLT of B019 in all subjects
MTD（Maximum tolerated dose） | Approximately 2 years
  Maximum tolerated dose

SECONDARY OUTCOMES:
The overall response rate (ORR) | Approximately 2 years
  Tumor response will be evaluated according to the Lugano 2014 criteria.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Zhujiang Hospital of Southern Medical University, Guangzhou
  - Jiangxi Cancer Hospital, Nanchang
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Xijing Hospital, Xi'an